CLINICAL TRIAL: NCT04383730
Title: Inhaled Sedation in COVID-19-related Acute Respiratory Distress Syndrome (ISCA): an International Research Data Study in the Recent Context of Widespread Disease Resulting From the 2019 (SARS-CoV2) Coronavirus Pandemics (COVID-19)
Acronym: ISCA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other); University Hospital Schleswig-Holstein (Other); Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Other Study IDs: ISCA Study
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Critically Illness; Sedation; Invasive Mechanical Ventilation; Acute Respiratory Distress Syndrome
Keywords: Mechanical ventilation; Acute Respiratory Distress Syndrome; Inhaled sedation; Intravenous sedation; Covid-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Usual practice of intravenous sedation: The choice of the intravenous sedative agent, including the type of and dosing of the agent, will be as per the treating clinicians at each center
  Interventions: Drug: Intravenous sedation
- Usual practice of inhaled sedation: The choice of the inhaled sedative agent, including the type of and dosing of the agent, will be as per the treating clinicians at each center.
  Interventions: Drug: Inhaled sedation

INTERVENTIONS:
Drug: Intravenous sedation — Patients will be included retrospectively in the study by local investigators at each participating center. As this is a non-interventional study, sedation practices will be those currently used as standard practices in participating centers, including both intravenous and inhaled sedation practices
  Groups: Usual practice of intravenous sedation
Drug: Inhaled sedation — Patients will be included retrospectively in the study by local investigators at each participating center. As this is a non-interventional study, sedation practices will be those currently used as standard practices in participating centers, including both intravenous and inhaled sedation practices
  Groups: Usual practice of inhaled sedation

SUMMARY:
The authors hypothesized that inhaled sedation, either with isoflurane or sevoflurane, might be associated with improved clinical outcomes in patients with COVID-19-related ARDS, compared to intravenous sedation.

The authors therefore designed the "Inhaled Sedation for COVID-19-related ARDS" (ISCA) non-interventional, observational, multicenter study of data collected from the patients' medical records in order to:

1. assess the efficacy of inhaled sedation in improving a composite outcome of mortality and time off the ventilator at 28 days in patients with COVID-19-related ARDS, in comparison to a control group receiving intravenous sedation (primary objective),
2. investigate the effects of inhaled sedation, compared to intravenous sedation, on lung function as assessed by gas exchange and physiologic measures in patients with COVID-19-related ARDS (secondary objective),
3. report sedation practice patterns in critically ill patients during the COVID-19 pandemics (secondary objective).

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is the most severe and lethal complication of COVID-19, and healthcare resource utilizations are currently being heavily challenged in most countries worldwide, with a high risk that some intensive care resources, such as the number of ventilators to allow management all patients, may be insufficient to face the current surge in ARDS cases. There is, therefore, an urgent need to evaluate candidate therapies that may impact clinical outcomes in patients with COVID-19-related ARDS and potentially be relevant to current public health issues, in accordance with the international efforts by the World Health Organization (WHO) (Global research on coronavirus disease) and most international public health organizations. Beyond the current efforts to find specific antiviral therapies or vaccines, improving supportive care and treatment options for patients with COVID-19-related ARDS, in accordance with up-to-date guidelines on the management of critically ill patients with COVID-19 (Surviving Sepsis Campaign: Guidelines on the Management of Critically Ill Adults with Coronavirus Disease 2019; The Australian and New Zealand Intensive Care Society (ANZICS) COVID-19 Guidelines; Recommandations d'experts SRLF-SFAR-SFMU-GFRUP-SPILF sur la prise en charge en réanimation des patients en période d'épidémie à SARS-CoV2), is of major importance.

Indeed, given the number of intensive care unit (ICU) patients for whom the question of sedation applies during the current COVID-19 outbreak, any sedation practice that would be associated with improved clinical outcomes could have significant economic and public health implications. In this perspective, the rationale supporting inhaled sedation with halogenated agents (such as isoflurane or sevoflurane) as a way to improve lung function, to decrease the inflammatory response, and to possibly improve patient outcome is strong.

The authors hypothesized that inhaled sedation, either with isoflurane or sevoflurane, might be associated with improved clinical outcomes in patients with COVID-19-related ARDS, compared to intravenous sedation. The authors, therefore, designed the "Inhaled Sedation for COVID-19-related ARDS" (ISCA) non-interventional, observational, multicenter study of data collected from the patients' medical records in order to :

1. assess the efficacy of inhaled sedation in improving a composite outcome of mortality and time off the ventilator at 28 days in patients with COVID-19-related ARDS, in comparison to a control group receiving intravenous sedation (primary objective),
2. investigate the effects of inhaled sedation, compared to intravenous sedation, on lung function as assessed by gas exchange and physiologic measures in patients with COVID-19-related ARDS (secondary objective),
3. report sedation practice patterns in critically ill patients during the COVID-19 pandemics (secondary objective).

This study will be performed in accordance with the Strengthening the Reporting of Observational studies in Epidemiology (STROBE) statement.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years old),
* Admitted to a participating ICU (or any other ICU-like setting that may be deployed as a result of the COVID-19 pandemics, such as in the operating room, post-anesthesia care unit, step-down unit or any COVID-19-specific unit set in response to the pandemics in a participating center),
* Requiring invasive mechanical ventilation,
* With suspected or confirmed COVID-19 on day 0.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in ICUrequiring invasive mechanical ventilation and suspected or confirmed COVID19
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of days off the ventilator (VFD28, for ventilator-free days), taking into account death as a competing event | Day 28 after inclusion
  Ventilator-free days to day 28 are defined as the number of days from the time of initiating unassisted breathing to day 28 after intubation, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a patient returns to assisted breathing and subsequently achieves unassisted breathing to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28. A period of assisted breathing lasting less than 24 hours and for the purpose of a surgical procedure will not count against the VFD calculation. If a patient was receiving assisted breathing at day 27 or died prior to day 28, VFDs will be zero. Patients transferred to another hospital or other health care facility will be followed to day 28 to assess this endpoint.

SECONDARY OUTCOMES:
All-cause mortality | Days 7, 14, and 28 after inclusion
  All-cause mortality
Ventilator-free days | Days 7 and 14 after inclusion
  Ventilator-free days to days 7 and 14 are defined as the number of days from the time of initiating unassisted breathing to day 7 and 14 after intubation, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to days 7 and 14 If a patient returns to assisted breathing and subsequently achieves unassisted breathing to days 7 and 14 , VFDs will be counted from the end of the last period of assisted breathing to days 7 and 14. A period of assisted breathing lasting less than 24 hours and for the purpose of a surgical procedure will not count against the VFD calculation. If a patient was receiving assisted breathing at day 6 or 13 or died prior to days 7 and 14, respectively,VFDs to days 7 and 14 will be zero. Patients transferred to another hospital or other health care facility will be followed to days 7 and 14 to assess this endpoint.
ICU-free days | Day 28 after inclusion
  Number of days alive and not in the ICU from inclusion to day 28
Duration of invasive mechanical ventilation | Day 28 after inclusion
  Total duration of controlled mechanical ventilation to day 28
Duration of controlled mechanical ventilation | Day 28 after inclusion
  Total duration of controlled mechanical ventilation to day 28
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  Arterial hypoxemia, as assessed by the partial pressure of arterial oxygen-to-fraction of inspired oxygen ratio (PaO2/FiO2)
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  Partial pressure of arterial carbon dioxide (PaCO2)
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  Inspiratory plateau pressure
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  Driving pressure
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  Mode of mechanical ventilation (assisted versus controlled)
Physiological measures of lung function | Days 1, 2, 3, 4, 5, 6, and 7 from inclusion
  If available, 100 ms occlusion pressure (P0.1), a marker of respiratory drive
Development of complications | Day 7 from inclusion
  Development of pneumothorax
Development of complications | Day 7 from inclusion
  Supraventricular tachycardia
Development of complications | Day 7 from inclusion
  New onset atrial fibrillation
Duration of vasopressor use | Day 28 after inclusion
  Total duration (in days) of vasopressor use
Duration of renal replacement therapy | Day 28 after inclusion
  Total duration (in days)of renal replacement therapy
Duration (in days) of any adjuvant therapies | Day 7 from inclusion
  Adjuvant therapies are defined as: prone position, recruitment maneuvers, inhaled nitric oxide, inhaled epoprostenol sodium, high frequency ventilation, ECMO, neuromuscular blockade
Duration of continuous neuromuscular blockade | Day 28 from inclusion
  Number of days with continuous neuromuscular blockade
Type of sedation practices | Day 28 from inclusion
  Sedation drug(s) used (name(s))
Duration of sedation practices | Day 28 from inclusion
  Number of days with sedation
Modalities of sedation practices | Day 28 from inclusion
  If inhaled sedation, device used to deliver it

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Jabaudon, Study Chair — University Hospital, Clermont-Ferrand
Locations (12):
- Beth Israel Deaconess Medical Center, Inc., Boston, Massachusetts, United States
- France (5):
  - CHU, Brest
  - CHU, Clermont-Ferrand
  - Centre Hospitalier, Dunkirk
  - Pitié-Salpêtrière Hospital - APHP, Paris
  - CH Privé de la Loire, Saint-Etienne
- Germany (3):
  - Universitätsklinikum, Bochum
  - University Medical Center Schleswig-Holstein, Kiel
  - Universitätsklinikum, Oldenburg
- Hospital Clínico Universitario de Valencia, Valencia, Spain
- Switzerland (2):
  - Cantonal Hospital, Münsterlingen
  - Universitätsspital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blondonnet R, Quinson A, Lambert C, Audard J, Godet T, Zhai R, Pereira B, Futier E, Bazin JE, Constantin JM, Jabaudon M. Use of volatile agents for sedation in the intensive care unit: A national survey in France. PLoS One. 2021 Apr 15;16(4):e0249889. doi: 10.1371/journal.pone.0249889. eCollection 2021. PMID 33857185